CLINICAL TRIAL: NCT03652519
Title: Influence of Different Rehabilitative Aerobic Exercise Programs on (Anti-) Inflammatory Immune Signalling, Cognitive Performance and Processing Skills in Persons With MS - A Randomized Controlled Trial
Brief Title: High-intensity Training and Its Effects on Neuroplasticity
Acronym: TRAINUVIMAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Valens (Other)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Principal Investigator, Jens Bansi, Sport Scientist and therapist, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BansiJ
Record Dates: First submitted 2018-08-14; First posted 2018-08-29 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Immune Signalling; Cognition; Health-related Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity Interval Training (HIIT) (Experimental): Participants of the HIIT group will exercise three times per week over a period of three weeks (inpatient rehabilitation) on a cycle ergometer. Exercise intensity will be regulated and heart rate controlled based on the achieved maximum heart rate (HRmax) assessed during the initial Cardiopulmonary Exercise Testing. Each exercise session will last 30 minutes and will be started and finalized with three minutes at low intensity (50% HRmax, warm-up / cool-down). During each exercise session, participants of the HIIT group will perform 5x one-and-a-half Minute high-intensive exercise bouts at 95-100% of their HRmax followed by active breaks of unloaded pedalling over 2 minutes with the aim to achieve 60% HRmax.
  Interventions: Behavioral: Exercise Training
- Moderate Continous Training (ST) (Active Comparator): Participants of the ST group will exercise three times per week over a period of three weeks (inpatient rehabilitation) on a cycle ergometer. Exercise intensity will be regulated and heart rate controlled based on the achieved maximum heart rate (HRmax) assessed during the initial Cardiopulmonary Exercise Testing. Each exercise session will last 30 minutes and will be started and finalized with three minutes at low intensity (50% HRmax, warm-up / cool-down). During each exercise session, participants of the ST group will exercise 30 minutes continuously at 65% of HRmax. This moderate continous training program represents the standard care at the local rehabilitation clinic.
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training — Treatment in both arms consists of specific of aerobic exercise training modalities. Exercise has become an efficient strategy within rehabilitative programs and is part of a goal-orientated multidisciplinary approach to improve disability and participation in persons with MS. Recently, short and exhaustive bouts of exercise have gained much attention as a promising option in supportive care in MS.

SUMMARY:
Regular physical activity is known to reduce the risk for some neurodegenerative disorders and their symptoms. Several studies have shown positive effects of therapeutic exercise interventions on motor- and cognitive function as well as psychosocial benefits in persons with multiple sclerosis (MS). To improve exercise recommendations, it is necessary to learn more about the underlying biological mechanisms. A reduction of inflammatory stress through physical exercise has been suspected as one key mechanism, mediating the positive effects of exercise in the context of MS (being a "classical" neuro-inflammatory disease). This randomized controlled trial aims to investigate the influence of two different rehabilitative endurance exercise programs (3x/week moderate vs. vigorous endurance exercise) on (1) (anti-)inflammatory immune signalling and (2) various aspects of participation.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of MS (according to the revised McDonald criteria 2010)
* Expanded Disability Status Scale 3.0 - 6.0
* Age > 21
* Relapsing remitting or secondary progressive MS
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Define drugs not allowed during the study or for specific periods of time prior to the administration of the test dose,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Tregs | Three weeks (day 0 to day 21)
  Proportion of regulatory T-cells with higher values indicating higher levels of Inflammation.

SECONDARY OUTCOMES:
Immune status | Three weeks (day 0 to day 21)
  Numbers and proportions of circulating immune cells associated with MS and exercise (Th17 cell, cytotoxic T-cells, naïve T-cells, memory T-cells, NK-cells, Monocytes) with higher values indicating higher levels of inflammation.
Soluble factors (cytokines, tryptophan metabolites, blood brain barrier markers) | Change from baseline (day 0) to directly after and 3-hours after the first exercise session (on day 0) and over 3-weeks (day 0 to day 21)
  Soluble factors that are known to be produced or secreted in response to (acute/chronic) exercise and are suspected to modify immune homeostasis and blood brain barrier function through their inflammatory and anti-inflammatory properties. (Tryptophan, Kynurenine, Kynurenine acid, Tumor Necrosis Factor-alpha (TNF-Alpha), Interferon-gamma (IFN-Gamma), Interleukin-6 (IL-6), Matrix-metalloproteinases-2 (MMP-2), Matrix-metalloproteinases-9 (MMP-9), Interleukin-10 (IL-10), Tumor Growth Factor-beta (TGF-beta), Interleukin-17 (IL-17) with higher values indicating higher levels of Inflammation.
Migratory Potential of peripheral mononuclear cells (PBMC) | Three weeks (day 0 to day 21)
  The migratory Potential of PBMC will be assessed by in situ zymography with higher values indicating higher Levels of Inflammation.
Endurance capacity | Three weeks (day 0 to day 21)
  Endurance capacity will be measured by peak oxygen consumption achieved in the cardiopulmonary exercise test. Higher values indicate better cardiorespiratory fitness.
Assessment of Motor and Processing Skills (AMPS) | Three weeks (day 0 to day 21)
  Processing skills of executive functions
Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) | Three weeks (day 0 to day 21)
  Cognitive Performance is assessed with the BICAMS This test battery involves three tests to assess the main cognitive domains vulnerable to MS: information processing speed, verbal and visual memory. The battery includes the Symbol Digit modalities Test (SDMT), Californian Verbal Learning Test-II (CVLT-II) and the Brief Visuospatial Memory Test revised (BVMT-R). Processing speed is the most relevant test and is assessed by the SDMT where the patients have 90s to voice numbers as rapidly as possible that were associated with target symbols within a grid printed at the top of a Stimulus page. The final score is the correct number of substitutions in 90 s, and scores ranges between 0 and 110. Higher scores indicating better cognition.
Fatigue Scale of Motor and cognitive function (FSMC) | Three weeks (day 0 to day 21)
  Changes of motor and cognitive fatigue on a 5-point Linkert-Scale. Max 50 Points for subsclaes, 100 Points for the Total score. Cut-off for fatigue is set for the total score at 43 and for the motoric and cognitive subscores at 22 with higher values participants being more fatigued.
Hospital Anxiety and Depression Scale (HADS) | Three weeks (day 0 to day 21
  Changes of anxiety and depression over three weeks training on a 4-point Linkert-Scale scored 0-3. Max 21 Points for each subsclae, cut off for anxiety and Depression are set at 7 Points higher values represent more anxiety and Depression.
Patient-Reported Outcome Measurement Information System (PROMIS) | Three weeks (day 0 to day 21)
  Changes of a 4-point Likert scale will provide information about the participants' healthcare-related quality of life with higher scores indicating better Quality of life.
Test battery of attention (TAP) | Three weeks (day 0 to day 21)
  Executive functions are assessed through the reaction time of the Go/No Go tasks of the TAP. Higher reaction times indicate better executive fuctionning.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bansi, PhD, Principal Investigator — Klinik Valens
Locations (1):
- Kliniken-Valens, Valens, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joisten N, Rademacher A, Warnke C, Proschinger S, Schenk A, Walzik D, Knoop A, Thevis M, Steffen F, Bittner S, Gonzenbach R, Kool J, Bloch W, Bansi J, Zimmer P. Exercise Diminishes Plasma Neurofilament Light Chain and Reroutes the Kynurenine Pathway in Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2021 Mar 29;8(3):e982. doi: 10.1212/NXI.0000000000000982. Print 2021 May. PMID 33782190
- [Derived] Joisten N, Rademacher A, Bloch W, Schenk A, Oberste M, Dalgas U, Langdon D, Caminada D, Purde MT, Gonzenbach R, Kool J, Zimmer P, Bansi J. Influence of different rehabilitative aerobic exercise programs on (anti-) inflammatory immune signalling, cognitive and functional capacity in persons with MS - study protocol of a randomized controlled trial. BMC Neurol. 2019 Mar 8;19(1):37. doi: 10.1186/s12883-019-1267-9. PMID 30849952